CLINICAL TRIAL: NCT03916991
Title: A Cross-over Study to Investigate the Effect of Hip-focused Neuromuscular Activation Exercise on Foot Posture and Neuromuscular Control
Brief Title: Effect of Hip-focused Neuromuscular Activation Exercise on Foot Posture and Neuromuscular Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, Associate Proffessor, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GO16542
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A cross-over study to investigate the effect of hip-focused neuromuscular activation exercise on foot posture and neuromuscular control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neuromuscular Exercise (Experimental): Neuromuscular Exercise
  Interventions: Other: Exercise
- Control (No Intervention): No intervention
- Sham Exercise (Sham Comparator): Sham Exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Hip focused Neuromuscular Activation Exercise
  Arms: Neuromuscular Exercise; Sham Exercise

SUMMARY:
This study planned to investigate the effect of hip-focused neuromuscular activation exercise on foot posture and neuromuscular control in symptomatic and asymptomatic participants. We will follow a cross-over study design to compare the effect of hip focused neuromuscular activation exercise or a sham exercise on foot posture and lower extremity biomechanics. Foot posture will be assessed by Navicular Drop Test (NDT), and lower extremity neuromuscular control will be assessed with Star Excursion Y-Balance Test (SEBT-Y) and Frontal Plane Projection Angle (FPPA) during single leg squat before and after the experiments. The results of this study may provide scientific knowledge for a kinetic chain approach during functional foot rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* To be included, participants should be between the ages of 18 and 45 years.

Exclusion Criteria:

* Participants will be excluded from this study if they have a history of lower body trauma or surgery, or positive trendelenburg sign and slump test.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-12 (Estimated); Primary Completion 2019-06-12 (Estimated); Study Completion 2019-07-12 (Estimated)

PRIMARY OUTCOMES:
Navicular Drop Test | 1 year
  Navicular Drop Test

SECONDARY OUTCOMES:
Star Excursion Y-Balance Test | 1 year
  Star Excursion Y-Balance Test
Frontal Plane Projection Angle | 1 year
  Frontal Plane Projection Angle

CONTACTS AND LOCATIONS:
Overall Officials: Elif Turgut, PhD, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No